CLINICAL TRIAL: NCT06980818
Title: Oral Microbiota Dysbiosis in Inflammatory Bowel Disease: a Cross-sectional Study Using Saliva as a Diagnostic Biomarker
Brief Title: Oral Microbiota Dysbiosis in IBD
Acronym: MIBD
Status: Active, not recruiting | Type: Observational
Sponsor: ULS Viseu Dão Lafões (Other)
Responsible Party: Principal Investigator, Rute Gomes, MD, ULS Viseu Dão Lafões
Other Study IDs: UIDP/04279/2020
Record Dates: First submitted 2025-03-26; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Disease (IBD); Dysbiosis
Keywords: IBD; Microbiome; Saliva
MeSH Terms: conditions — Inflammatory Bowel Diseases; Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples Without DNA — Biospecimens will be saliva and biofilm samples from patients with IBD and healthy controls. The collected biological samples will be analyzed at SalivaTec using molecular biology and immunology approaches, no DNA will be extracted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IBD patients: Patients with Crohn's disease or ulcerative colitis
  Interventions: Other: No intervention
- Control group: Age-matched unrelated healthy individuals
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will take place.

SUMMARY:
This study aims to provide new insights into oral microbiota dysbiosis and IBD. Given the strong association between oral health, microbiome composition, and IBD, all participants will undergo an oral evaluation program conducted by dentists from the Faculty of Dentistry at Universidade Católica Portuguesa (UCP). This program will facilitate the characterization of oral health and its correlation with IBD status.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) can impact the entire gastrointestinal tract, from the oral cavity to the anal region, particularly in Crohn's disease, making oral conditions recognized as extraintestinal manifestations. A clear link exists between the severity of IBD and disruptions in the oral microbial community. These extraintestinal manifestations often appear as various lesions in the oral cavity, including aphthous ulcers, recurrent aphthous stomatitis (RAS), granulomas, gingival inflammation, periodontitis, and angular cheilitis. The severity and prevalence of these conditions correlate with the extent of intestinal inflammation.

Research has shown that the intake of excessive amount of imbalanced oral bacteria-such as those resulting from periodontitis-can compromise the gut barrier, leading to impaired gut function, alterations in intestinal microbiota, and immune dysfunction. IBD patients are more susceptible to severe forms of periodontitis compared to individuals with periodontal disease without chronic inflammation. They exhibit greater probing depths, increased plaque levels, bleeding on probing, calculus buildup, and more significant clinical attachment loss (CAL). This bidirectional relationship suggests that while IBD patients are more prone to periodontitis, periodontitis itself may also elevate the risk of developing IBD. The oral cavity hosts over 250 bacterial species, including known periodontal pathogens such as Tannerella forsythia, Streptococcus mutans, Aggregatibacter actinomycetemcomitans, and Porphyromonas gingivalis. When these bacteria exceed normal levels, they can enter the bloodstream through mechanical actions like brushing or dental procedures. Once in circulation, they invade and colonize immune cells such as macrophages and dendritic cells, ultimately reaching and spreading throughout the highly vascularized intestinal tract.

Saliva plays a crucial role in this process, acting as a transporter that facilitates bacterial survival by protecting them from stomach acid through its composition of proteins, lipids, water, and mucins.

While the gut microbiome's role in IBD has been widely studied, limited research has explored the contribution of the oral microbiome to the development of this disease and the associated oral conditions in IBD patients.

Primary Objective:

- Assess the dysbiosis of the oral microbiome in patients with IBD compared to healthy controls.

Secondary Objectives:

* Identify key bacterial species in the salivary microbiome that differentiate IBD patients from healthy individuals.
* Evaluate correlations between oral microbiota composition and clinical parameters (e.g., duration of disease, tobacco use, disease activity, presence of oral symptoms). This will be a cross-sectional observational study designed to assess the dysbiosis of the oral microbiome in patients with IBD compared to healthy controls. The study will involve only one point of evaluation, focusing on saliva samples for microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old and diagnosis of IBD according to established criteria

Exclusion Criteria:

* Recent history of antibiotic treatment (within the preceding month), proton pump inhibitors or non-steroidal anti-inflammatory drugs were exclusion criteria for both patients and controls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who met the inclusion criteria were followed in the IBD consultation at the Gastroenterology Department of ULS Viseu Dão-Lafões.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral microbiome characterization | 3 years
  Assess the dysbiosis of the oral microbiome in patients with IBD compared to healthy controls.

SECONDARY OUTCOMES:
Bacterial species characterization in IBD | 3 years
  Identify key bacterial species in the salivary microbiome that differentiate IBD patients from healthy individuals.
Does oral microbiota correlates with disease activity? | 3 years
  Evaluate correlations between oral microbiota composition and clinical parameters (e.g., duration of disease, tobacco use, disease activity, presence of oral symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Paula Ministro, MD, Study Director — ULS Viseu Dão Lafões
Locations (1):
- ULS Viseu Dão-Lafões, Viseu, Viseu District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chandan JS, Thomas T. The impact of inflammatory bowel disease on oral health. Br Dent J. 2017 Apr 7;222(7):549-553. doi: 10.1038/sj.bdj.2017.318. PMID 28387295